CLINICAL TRIAL: NCT01206595
Title: A Phase 2, Multicenter, Randomized, Double Blind, Dose Escalating/ De-Escalating Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of Sustained Release Encapsulated Bupivacaine (SKY0402) Administered as a Nerve Block in the Management of Postoperative Pain in Subjects Undergoing Bunionectomy
Brief Title: Safety, Efficacy, and Pharmacokinetics of SKY0402 Administered as a Nerve Block in Subjects Undergoing Bunionectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SKY0402-C-203
Record Dates: First submitted 2010-09-19; First posted 2010-09-22 (Estimated); Results first posted 2012-05-15 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Postoperative Pain
Keywords: Postoperative Pain; Bunionectomy; Analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SKY0402 (Active Comparator): Low-dose (175 mg), low-mid dose( 225 mg), and mid-dose (350 mg)
  Interventions: Drug: SKY0402
- Bupivacaine HCl (Active Comparator): Marcaine with epinephrine 1:200,000 is the reference-listed drug for bupivacaine and contains the same active, local anesthetic as SKY0402
  Interventions: Drug: Bupivacaine HCl

INTERVENTIONS:
Drug: SKY0402 — Single dose of SKY0402 administered as a nerve block
  Arms: SKY0402
Drug: Bupivacaine HCl — Single dose of 125 mg administered as a nerve block
  Arms: Bupivacaine HCl

SUMMARY:
The primary objective of this study was to determine the appropriate dose of SKY0402 administered as a nerve block for the management of postoperative pain following bunionectomy.

DETAILED DESCRIPTION:
This Phase 2, multicenter, randomized, double blind, dose escalating/de-escalating study evaluated the safety, efficacy, and pharmacokinetics of a single dose of SKY0402 compared to a single 125 mg dose of bupivacaine HCl for the treatment of postoperative pain in subjects undergoing bunionectomy.

Up to 88 subjects were to be randomized in five consecutive cohorts. The dose of bupivacaine HCl (125 mg) was to remain constant for all cohorts. After completion of Cohort 1, the decision to increase or decrease the dose of SKY0402 was made by a Cohort Data Review Committee following a review of pharmacokinetic, safety, and selected efficacy data from the previous cohort.

Study drug was to be administered as an ankle block, with or without a tourniquet, between 1 hour before the induction of general anesthesia and 20 minutes before the end of general anesthesia. The ankle block procedure consisted of five injections via three skin entries targeting the following nerves: posterior tibial, sural, deep peroneal, superficial peroneal, and saphenous.

The use of intravenous fentanyl during general anesthesia was permitted, but was not to exceed 250 micrograms. The intraoperative use of morphine was prohibited. Postoperatively, subjects had access to both opioid and non-opioid supplemental pain medication under general guidelines. Blood samples for the determination of plasma bupivacaine concentrations were obtained at Baseline and at specified time points through 96 hours.

ELIGIBILITY:
Inclusion Criteria:

Subjects were eligible for enrollment if they met the following criteria:

1. Males and females ≥18 years of age at the Screening Visit. NOTE: Eligible females were postmenopausal or surgically sterile, or, if of child bearing potential, were not pregnant or nursing, and they agreed to not become pregnant during the study by using acceptable means of contraception for at least 1 month before and 1 month after dosing, including any of the following: hormonal contraceptives (oral, injectable, implantable), effective barrier methods (e.g., condoms with spermicide), intrauterine device (IUD), lifestyle with a personal choice of abstinence, non-heterosexual lifestyle, or in a strictly monogamous relationship with a partner who has had a vasectomy.
2. Scheduled to undergo a primary unilateral first metatarsal bunionectomy repair under general anesthesia, with or without internal fixation.

   NOTE: For the purpose of this protocol, all surgical procedures involving osteotomy of the first metatarsal (significant bone resection, excision, surgical fracture, etc.) or fusion of the first metatarsal phalangeal joint were considered qualified procedures, whether or not performed specifically to repair a bunion (hallus valgus deformity). Surgical techniques accompanied by minimal bone excision (e.g. cheilectomy) or procedures limited to soft tissue repair were not eligible for this study.
3. American Society of Anesthesiology (ASA) Physical Class 1 or 2.
4. Able and willing to comply with all study visits and procedures.
5. Capable of speaking and understanding the local language sufficiently to provide responses to pain assessment scales.
6. Willing and capable of providing written informed consent.

Exclusion Criteria:

Subjects were excluded from the study if they met any of the following criteria:

1. Clinically significant electrocardiogram (ECG) abnormalities at Screening or on Day 1 (before dosing).
2. Albumin and/or alpha 1 acid glycoprotein (AAG) below normal levels.
3. Current or historical evidence of any clinically significant disease or condition that, in the opinion of the Investigator, might have increased the risk of surgery or complicated the subject's postoperative course.
4. Opioid medication usage during the 7 day period preceding the administration of study drug.
5. Current medical conditions that could have required treatment with analgesic medications in the postoperative period for pain that was not surgically related (e.g., rheumatoid arthritis).
6. Body mass index >30 kg/m^2.
7. Body weight less than 60 kilograms.
8. History of hypersensitivity or idiosyncratic reaction to amide type local anesthetic agents.
9. History of hypersensitivity, idiosyncratic reactions, and other contraindications to the pain control agents (opioid or non-opioid) anticipated to be used postoperatively. These contraindications may have included the following: angioedema and bronchospastic reactivity to non-steroidal anti-inflammatory drug (NSAID), peptic ulcer (active within the last 3 months), or hepatic or renal insufficiency.
10. Coagulation disorders or ongoing anticoagulation treatment.
11. Administration of an investigational drug within 30 days or 5 half lives (of elimination), whichever was longer, prior to study drug administration.
12. Suspected or known history of substance abuse and/or alcoholism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2005-03; Primary Completion 2006-03 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kay Warnott, RN, ACNP, Study Director — Parica Pharmaceuticals, Inc.

RESULTS

PARTICIPANT FLOW:
Groups:
- SKY0402: Low-dose, low-mid dose, and mid-dose
Period: Overall Study
Arm/Group | SKY0402 | Bupivacaine HCl
Started | 38 | 20
Completed | 38 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SKY0402 | Bupivacaine HCl | Total
Number analyzed (Participants) | 38 | 20 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 15 | 44
  >=65 years | 9 | 5 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (14.04) | 55.7 (14.22) | 54.8 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 18 | 48
  Male | 8 | 2 | 10
Region of Enrollment [Number; unit: participants]
  Australia | 3 | 5 | 8
  Belgium | 29 | 12 | 41
  United Kingdom | 3 | 2 | 5
  Netherlands | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Time to First Use of Supplemental Pain Medication Postoperatively for Surgical Pain
Description: The primary efficacy endpoint was the time to first use of supplemental pain medication (opioid or non-opioid) postoperatively for surgical pain.
Time Frame: Through 96 hours postdose
Measure: Median (Inter-Quartile Range); unit: hours
Groups:
- Bupivacaine HCl: A single dose of bupivacaine HCl 125 mg was administered intraoperatively by local infiltration.
- SKY0402 Low Dose (175 mg): A single dose of SKY0402 Low Dose (175 mg) was administered intraoperatively by local infiltration.
- SKY0402 Low-Mid Dose (225 mg): A single dose of SKY0402 low-mid dose (225 mg) was administered intraoperatively by local infiltration.
- SKY0402 Mid Dose (350 mg): A single dose of SKY0402 mid dose (350 mg) was administered intraoperatively by local infiltration.
Arm/Group | Bupivacaine HCl | SKY0402 Low Dose (175 mg) | SKY0402 Low-Mid Dose (225 mg) | SKY0402 Mid Dose (350 mg)
Number analyzed (Participants) | 20 | 12 | 12 | 14
hours | 9.4 [6.1 to 11.2] | 1.9 [0.3 to 9.0] | 1.2 [0.6 to 5.4] | 2.4 [0.3 to 8.3]

2. Secondary Outcome: Number of Patients With Adverse Events
Description: All adverse events were to be recorded from the time of dosing through Day 8. Serious adverse events (SAEs) were to be recorded through Day 30.
Time Frame: Through 30 days postdose
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | SKY0402 | Bupivacaine HCl
Serious Adverse Events (participants affected / at risk) | 1/38 | 0/20
Other Adverse Events (participants affected / at risk) | 15/38 | 6/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SKY0402 (N=38) | Bupivacaine HCl (N=20)
Immobiliaztion prolonged (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SKY0402 (N=38) | Bupivacaine HCl (N=20)
Bradycardia (Cardiac disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 9 | 3
Vomiting (Gastrointestinal disorders) | 3 | 0
Headache (Nervous system disorders) | 2 | 0
Hypotension (Vascular disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No